CLINICAL TRIAL: NCT02361138
Title: Pharmacokinetics, Pharmacodynamics, Safety and Tolerability Study Following Multiple Dose of SHR3824 in Healthy Subjects
Brief Title: The PK/PD Study of Multiple Dose of SHR3824 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR3824-102
Record Dates: First submitted 2015-02-01; First posted 2015-02-11 (Estimated); Last update posted 2015-02-11 (Estimated); Status verified 2014-12

CONDITIONS: Type 2 Diabetes
Keywords: SHR3824 Type 2 diabetes mellitus SGLT2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — henagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Cohort SHR3824/Placebo 1.25 mg (Experimental): SHR3824 1.25 mg/day or placebo for 10 days.
  Interventions: Drug: SHR3824; Drug: Placebo
- Cohort SHR3824/Placebo 2.5 mg (Experimental): SHR3824 2.5 mg/day or placebo for 10 days. The actual dose (mg) level selected for each cohort may be modified based on evaluation of preliminary safety, pharmacokinetic and pharmacodynamic data from previous cohort.
  Interventions: Drug: SHR3824; Drug: Placebo
- Cohort SHR3824/Placebo 5 mg (Experimental): SHR3824 5 mg/day or placebo for 10 days. The actual dose (mg) level selected for each cohort may be modified based on evaluation of preliminary safety, pharmacokinetic and pharmacodynamic data from previous cohort.
  Interventions: Drug: SHR3824; Drug: Placebo
- Cohort SHR3824/Placebo 10 mg (Experimental): SHR3824 10 mg/day or placebo for 10 days. The actual dose (mg) level selected for each cohort may be modified based on evaluation of preliminary safety, pharmacokinetic and pharmacodynamic data from previous cohort.
  Interventions: Drug: SHR3824; Drug: Placebo
- Cohort SHR3824/Placebo 25 mg (Experimental): SHR3824 25 mg/day or placebo for 10 days. The actual dose (mg) level selected for each cohort may be modified based on evaluation of preliminary safety, pharmacokinetic and pharmacodynamic data from previous cohort.
  Interventions: Drug: SHR3824; Drug: Placebo
- Cohort SHR3824/Placebo 100mg (Experimental): SHR3824 100 mg/day or placebo for 10 days. The actual dose (mg) level selected for each cohort may be modified based on evaluation of preliminary safety, pharmacokinetic and pharmacodynamic data from previous cohort.
  Interventions: Drug: SHR3824; Drug: Placebo

INTERVENTIONS:
Drug: SHR3824
  Other Names: Henagliflozin
Drug: Placebo

SUMMARY:
SHR3824 is a novel inhibitor of renal sodium-glucose cotransporter 2, allows an insulin-independent approach to improve type 2 diabetes hyperglycemia. In this multiple-dose study the investigators evaluated the safety, tolerability and PK/PD profiles of SHR3824 in healthy subjects.

ELIGIBILITY:
Inclusion criteria:

* Chinese male and female subjects aged 18 to 45 years.
* BMI:18 -25 kg/m2.
* Healthy according to medical history, physical examination findings, 12-lead ECG findings, and clinical laboratory evaluations.

Exclusion criteria:

* History of or current clinically significant medical illness as determined by the Investigator.
* History of clinically significant allergies, especially known hypersensitivity or intolerance to lactose.
* Pregnancy or breastfeeding . Significant acute or chronic medical illness, including renal impairment, or recent surgery.
* Donation of blood or plasma within the 4 weeks prior to the start of the study or acceptance of blood transfusion within 8 weeks.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2013-12; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
AUC(Area under the curve) of SHR3824. | day1 and day11 to day 13.
Cmax(the maximum concentration) of SHR3824. | day1 and day11 to day 13.
Tmax(the time reaching maximum concentration) of SHR3824. | day1 and day11 to day 13.
Halflife of SHR3824. | day1 and day11 to day 13.
CL/F of SHR3824. | day1 and day11 to day 13.
V/F of SHR3824. | day1 and day11 to day 13.
Accumulation ratio of SHR3824 | Up to day 13.
Urine glucose concentration of SHR3824. | day1 and day11
Plasma glucose concentration of SHR3824. | day1 and day11

SECONDARY OUTCOMES:
Adverse events, vital signs, physical exams , ECG, clinical labs | Days -14 to -1, 0, 13.
Serum creatinine | Days -14 to -1, 0, 2, 9, 13.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Xuhui Central Hospital, Shanghai, Shanghai Municipality, China